CLINICAL TRIAL: NCT05059691
Title: Three-Dimensional Fluoroscopic Guidance During Transbronchial Cryobiopsy, a Prospective Pilot Study
Brief Title: Three-Dimensional Fluoroscopic Guidance During Transbronchial Cryobiopsy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1174; NCI-2021-08947 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1174 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-10; First posted 2021-09-28 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (transbronchial cryobiopsy): Patients undergo transbronchial cryobiopsy guided by three-dimensional fluoroscopy. Patients' medical records are also reviewed.
  Interventions: Other: Electronic Health Record Review; Procedure: Transbronchial Cryobiopsy Guided by Three-Dimensional Fluoroscopy

INTERVENTIONS:
Other: Electronic Health Record Review — Review of medical records
Procedure: Transbronchial Cryobiopsy Guided by Three-Dimensional Fluoroscopy — Undergo transbronchial cryobiopsy guided by three-dimensional fluoroscopy

SUMMARY:
This study assesses the effectiveness of transbronchial cryobiopsy guided by 3-dimensional fluoroscopy. Transbronchial cryobiopsy is a procedure to collect lung tissue. The main side effect seen after a transbronchial cryobiopsy is pneumothorax (air leaking out of the lung, which may cause a completely or partially collapsed lung). The standard imaging scans used during this procedure are 2-dimensional (like a photo), which can make it difficult for the doctor to know exactly where the biopsy tool is during the procedure. If the exact location of the device is not clear, a patient can be at a higher risk of pneumothorax. Using a 3-dimensional imaging technique may help to decrease the risk of pneumothorax during transbronchial cryobiopsy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if transbronchial cryobiopsy guided by three-dimensional fluoroscopy reduces the incidence of pneumothorax up to 72 hours after transbronchial cryobiopsy.

SECONDARY OBJECTIVE:

I. To describe outcomes of cryobiopsy, need for interventions related to transbronchial cryobiopsy, radiation dose, and any complications or adverse events after transbronchial cryobiopsy guided by three-dimensional fluoroscopy.

OUTLINE:

Patients undergo transbronchial cryobiopsy guided by three-dimensional fluoroscopy. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Presence of an intraparenchymal lung lesion for which cryobiopsy is deemed the most appropriate method of biopsy
* Ability to provide informed consent

Exclusion Criteria:

* Acute respiratory failure (defined as oxygen requirement > 4 L/min by nasal cannula above baseline, or need for any intervention to support ventilation and/or gas exchange for any duration, including invasive and non-invasive positive pressure ventilation, high-flow therapy, non-rebreather mask, or Venturi mask)
* Intensive care unit (ICU) admission
* Forced vital capacity (FVC) < 50% or diffusing capacity of the lung for carbon monoxide (CO) (DLCO) < 35% (if pulmonary function tests are available)
* Known or suspected pulmonary hypertension (defined as elevated right ventricular systolic pressure on echocardiogram, if available)
* Acute renal failure or chronic kidney disease
* Platelets < 100,000/uL
* International normalized ratio (INR) > 1.5
* Use of anticoagulant therapy that cannot be held for 2 days
* Use of antiplatelet therapy (other than baby aspirin) that cannot be held for 5 days
* Any bleeding diathesis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with presence of an intraparenchymal lung lesion for which cryobiopsy is deemed the most appropriate method of biopsy
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Incidence of pneumothorax | Up to 72 hours after cryobiopsy
  The proportion of patients developing pneumothorax will be compared with the proportion in the historical control (i.e., 20%) using two-sided binomial test. A p-value of less than 0.05 will indicate a statistical significance. The proportion of patients identified as developing pneumothorax and its exact 95% confidence interval will be estimated. Poisson regression model will be used to estimate the incidence of pneumothorax accounting for the number of biopsy sites.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce F Sabath, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org